CLINICAL TRIAL: NCT04378595
Title: Assessing Pediatric Food Insecurity During the COVID-19 Pandemic in Austin Federally Qualified Health Centers
Brief Title: Assessing Pediatric Food Insecurity During the COVID-19 Pandemic in Austin
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Texas at Austin (Other)
Responsible Party: Principal Investigator, Steven Abrams, Professor, University of Texas at Austin
Other Study IDs: 2020-004-0019
Record Dates: First submitted 2020-05-05; First posted 2020-05-07 (Actual); Last update posted 2020-05-08 (Actual); Status verified 2020-05

CONDITIONS: Food Insecurity
Keywords: food insecurity; COVID-19; pandemic
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- During Pandemic: During Pandemic: The investigators will query the parent/guardian with the 2-question food insecurity validated tool during their regular appointment, either in person or on the phone/telehealth. If a positive response is given, the investigators will ask if the food insecurity began or worsened during the pandemic in the past 1 to 2 months.
  Interventions: Other: During COVID-19 Pandemic
- Post-Pandemic: Post-Pandemic: The investigators will query the parent/guardian with the 2-question food insecurity validated tool during their regular appointment, either in person or on the phone/telehealth. The investigators will assess if food insecurity has stopped or lessened after the pandemic.
  Interventions: Other: After COVID-19 Pandemic

INTERVENTIONS:
Other: During COVID-19 Pandemic — Assessing status of food insecurity during the COVID-19 pandemic
  Groups: During Pandemic
Other: After COVID-19 Pandemic — Assessing status of food insecurity after the COVID-19 pandemic
  Groups: Post-Pandemic

SUMMARY:
The investigators suspect that the current COVID-19 pandemic may be associated with a high level of unsuspected food insecurity among lower income Austin families who receive their health care at a Federally Qualified Health Center (FQHC). Pediatricians will ask families about food insecurity as part of standard of care in order to assess if food insecurity has begun or worsened during the pandemic.

DETAILED DESCRIPTION:
According to previous studies, 21-23% of lower income families experience food insecurity, a position of uncertainty about their ability to afford food or omitting meals for financial reasons. Food insecurity in a family is detrimental to a child's mental and physical health, and poses a risk to his/her development. Food insecurity prevalence has also been reported higher than the state level prevalence in households impacted by disasters. It is therefore reasonable to hypothesize that the unprecedented global COVID-19 pandemic has increased the frequency of food insecurity among lower income families. However, no data are known about the current incidence of food insecurity during a pandemic with quarantine procedures in place. This knowledge will also add background for future studies on the effects of acute on chronic food insecurity on low-income families facing similar adversities such as this epidemic.

A 2-question tool has been validated to evaluate the presence of food insecurity. An affirmative response to either question has been reported to yield a sensitivity of 97% and specificity of 83-86%. Screening for basic needs may open a sensitive discussion about economic difficulties associated with the adverse health outcomes previously discussed. While this tool is a current standard of care as recommended by the American Academy of Pediatrics, it is often not utilized in medical visits to a primary care provider whether for routine well child care or for sick visits. During the study period, pediatricians at two FQHC clinics will make a concentrated effort to ask these 2 screening questions in order to collect data on the prevalence and magnitude of challenges of food insecurity at this time.

Although the investigators are seeking to evaluate the current standard of care, they may want to share our findings in order to provide a foundation for more generalizable research.

The investigators will seek to take a random sampling of 500 pediatric patients (250 each from 2 CommUnity Care clinics) and query the parent/guardian with the 2-question food insecurity tool during their regular appointment, either in person or on the phone/telehealth. The pediatricians (Co-Inv) will ask the questions and record the data.

2-questions to assess food insecurity as recommended by the American Academy of Pediatrics:

1. "We worried whether our food would run out before we got money to buy more." Was that often true, sometimes true, or never true for your household in the last 12 months?
2. "The food we bought just didn't last, and we didn't have money to get more." Was that often true, sometimes true, or never true for your household in the last 12 months? A response of "often true" or "sometimes true" to either question = positive screen for Food Insecurity.

The investigators will also ask the same 2 questions in the framework of "…in the last 1-2 months" to assess how the current situation has affected their immediate concerns. If the parent/guardian response with a positive screen for food insecurity, the pediatrician will refer the families to available community resources as is the usual standard of care.

The investigators will not record any identifiable information. This is not a longitudinal study. In 4-6 months the investigators will repeat this procedure with another, different random sampling of 500 patients to assess any long lasting effects of the COVID-19 pandemic or to determine if the immediate food crisis due to the pandemic has passed. The investigators requested a waiver of consent for this project.

ELIGIBILITY:
Inclusion Criteria:

* Any parent/caregiver of a pediatric patient being seen at the 2 specified CommUnity Care centers

Exclusion Criteria:

* Not at 2 specified CommUnity Care centers under care of researchers

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Parent/Caregiver of pediatric patients at 2 specified CommUnity Care centers (Rundberg clinic and Southeast Health and Wellness Clinic)
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2020-04-10 (Actual); Primary Completion 2020-12-30 (Estimated); Study Completion 2021-07-30 (Estimated)

PRIMARY OUTCOMES:
Food Insecurity Score | Up to 1 year
  2-questions to assess food insecurity as recommended by the American Academy of Pediatrics:
  1. "We worried whether our food would run out before we got money to buy more." Was that often true, sometimes true, or never true for your household in the last 12 months?
  2. "The food we bought just didn't last, and we didn't have money to get more." Was that often true, sometimes true, or never true for your household in the last 12 months? A response of "often true" or "sometimes true" to either question = positive screen for Food Insecurity.
  The investigators will also ask the same 2 questions in the framework of "…in the last 1-2 months" to assess how the current situation has affected their immediate concerns, assessing if their food insecurity has begun or worsened during the pandemic.

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Dell Medical School, Austin, Texas
  - CommUnity Care Clinic - Southeast Health and Wellness Clinic, Austin, Texas
  - CommUnity Care Clinic - Rundberg, Austin, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Rose-Jacobs R, Black MM, Casey PH, Cook JT, Cutts DB, Chilton M, Heeren T, Levenson SM, Meyers AF, Frank DA. Household food insecurity: associations with at-risk infant and toddler development. Pediatrics. 2008 Jan;121(1):65-72. doi: 10.1542/peds.2006-3717. PMID 18166558
- [Background] Hager ER, Quigg AM, Black MM, Coleman SM, Heeren T, Rose-Jacobs R, Cook JT, Ettinger de Cuba SA, Casey PH, Chilton M, Cutts DB, Meyers AF, Frank DA. Development and validity of a 2-item screen to identify families at risk for food insecurity. Pediatrics. 2010 Jul;126(1):e26-32. doi: 10.1542/peds.2009-3146. PMID 20595453
- [Background] Clay LA, Ross AD. Factors Associated with Food Insecurity Following Hurricane Harvey in Texas. Int J Environ Res Public Health. 2020 Jan 25;17(3):762. doi: 10.3390/ijerph17030762. PMID 31991735
- [Background] Gattu RK, Paik G, Wang Y, Ray P, Lichenstein R, Black MM. The Hunger Vital Sign Identifies Household Food Insecurity among Children in Emergency Departments and Primary Care. Children (Basel). 2019 Oct 2;6(10):107. doi: 10.3390/children6100107. PMID 31581751
- [Derived] Abrams SA, Avalos A, Gray M, Hawthorne KM. High Level of Food Insecurity among Families with Children Seeking Routine Care at Federally Qualified Health Centers during the Coronavirus Disease 2019 Pandemic. J Pediatr X. 2020 Fall;4:100044. doi: 10.1016/j.ympdx.2020.100044. Epub 2020 Jun 22. PMID 32864604
- See also: AAP Tool Kit for Food Insecurity — http://frac.org/aaptoolkit